## Cover letter

Official Title: Evaluation of the Clinical and Growth-related effects of Probiotics in Preterm Infant: A Randomized, Placebo Controlled Clinical Trial.

NCT number: not assigned yet

Date: 10 May 2023

## **CONSENT FORM**

<u>Title: Evaluation of the Clinical and Growth-related effects of Probiotics in Preterm Infant: A</u>

<u>Randomized, Placebo Controlled Clinical Trial.</u>

| • Name of PI: Dr. Imran Masood | Field Supervisor: Dr. Imran Qaiser • | Co-investigator: |
|---|---|---|
| Madiha | | |

| Participant name |
|---------------------|
| Screening ID number |

## STATEMENT OF PERSON GIVING CONSENT:

- 1. I confirm that I have read the information sheet for the study above, or it has been explained to me in a language I am familiar with.
- 2. I have spoken with the doctor to my satisfaction, and I've had the chance to ask any questions
- 3. I understand that participation of my child is completely voluntary. I have received sufficient information about the research study to decide whether I want to take part.
- 4. I understand that I have the freedom to withdraw at any time, without giving any explanation and that medical care or legal rights of my child will not be compromised.
- 5. I am aware that I will receive a copy of this consent form and the information sheet to keep for my records.
- 6. I understand that the study staff might look into my child's medical records and I give them permission to do so.
- 7. I am aware that my child's data will be available to the public with all personal information omitted.
- 8. I agree to a copy of this consent form which includes my child's personal information being made available to Department of Pharmacy Practice, Faculty of Pharmacy, The Islamia University of Bahawalpur for the purpose of monitoring only.

| 9. I consent to my child's participation in the study m | nentioned above. |
|---|---|
| Name of patient's parent/authorized guardian | Signature/ thumbprint |
| Date | |
| STATEMENT OF PERSON OBTAINING INFORMED CO<br>I have provided a detailed explanation of this resear<br>benefits to make an informed decision. | |
| Name | Date |